CLINICAL TRIAL: NCT07234071
Title: The Effectiveness of Manual Therapy Combined With Functional Magnetic Stimulation in Individuals With Lumbar Radiculopathy Due to Lumbar Disc Herniation: A Randomized Controlled Trial
Brief Title: Manual Therapy Combined With Functional Magnetic Stimulation for Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Assistant Professor of Physiotherapy, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-16/2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Lumbar Disc Herniation With Radiculopathy
Keywords: Lumbar Radiculopathy; Low Back Pain; Root Compression, Neuropathic Pain; Acute Radicular Pain
MeSH Terms: conditions — Radiculopathy; Low Back Pain; Neuralgia | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: A single-assessor-blind randomized controlled trial will be conducted over three weeks in forty adults with lumbar radiculopathy due to lumbar disc herniation. Participants will be randomly allocated 1:1 (n = 20 per group) to either: (1) manual therapy (neurodynamic mobilization) combined with Functional Magnetic Stimulation (FMS), or (2) the same manual therapy protocol without FMS. Both groups will complete ten treatment sessions during the three-week period. Clinical assessments-including pain intensity (Numeric Pain Rating Scale), functional disability (Roland-Morris Disability Questionnaire), straight leg raise (SLR) angle measured with goniometry, and neuropathic symptoms (S-LANSS, Greek)-will be obtained at baseline and at the end of the three-week intervention.
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor) A masked assessor will conduct the measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy and Functional Magnetic Stimulation (Experimental): Participants allocated to this group will receive 10 sessions of manual therapy with Functional Magnetic Stimulation
  Interventions: Other: Combined manual therapy and Functional Magnetic Stimulation
- Manual Therapy without Functional Magnetic Stimulation (Active Comparator): Participants allocated to this group will receive 10 sessions of a Manual Therapy without Functional Magnetic Stimulation.
  Interventions: Other: Manual Therapy without Functional Magnetic Stimulation

INTERVENTIONS:
Other: Combined manual therapy and Functional Magnetic Stimulation — Participants allocated to this group will receive a combined program consisting of neurodynamic manual therapy and Functional Magnetic Stimulation (FMS). The manual therapy protocol includes symptom-guided spinal mobilization with leg movement and standardized sciatic nerve mobilization techniques. FMS will be applied using a high-intensity magnetic stimulator targeting the lumbosacral nerve roots and the sciatic nerve pathway. A total of 10 treatment sessions will be administered over a 3-week period.
  Arms: Manual Therapy and Functional Magnetic Stimulation
Other: Manual Therapy without Functional Magnetic Stimulation — Participants in this group will receive the same neurodynamic manual therapy protocol as the experimental group, including symptom-guided spinal mobilization with leg movement and sciatic nerve mobilization techniques. However, they will not receive Functional Magnetic Stimulation (FMS). A total of 10 treatment sessions will be administered over the 3-week intervention period.
  Arms: Manual Therapy without Functional Magnetic Stimulation

SUMMARY:
This randomized clinical trial will evaluate whether adding Functional Magnetic Stimulation (FMS) to manual therapy (neurodynamic mobilization) improves clinical outcomes in adults with lumbar radiculopathy caused by lumbar disc herniation. Forty participants will be randomly assigned to two groups: an intervention group receiving manual therapy combined with FMS and a control group receiving manual therapy alone. All participants will complete a three-week physiotherapy program consisting of ten treatment sessions. Outcomes will be assessed at baseline and at the end of the three-week intervention period. Primary outcomes include pain intensity (Numeric Pain Rating Scale, NPRS), functional disability (Roland-Morris Disability Questionnaire, RMDQ), straight leg raise (SLR) range of motion measured with goniometry, and neuropathic symptom characteristics (S-LANSS, Greek). The study aims to determine whether the addition of FMS produces superior clinical improvements compared with manual therapy alone.

DETAILED DESCRIPTION:
Background: Lumbar disc herniation with radiculopathy is a common musculoskeletal and neurological condition caused by compression or irritation of the lumbar nerve roots, often leading to radiating leg pain, paresthesia, and movement limitation. Neural (neurodynamic) mobilization is a manual physiotherapy technique aiming to restore the mechanical and physiological interface between neural tissues and their surrounding structures, thereby improving nerve mobility and reducing mechanosensitivity. Functional Magnetic Stimulation (FMS) is a non-invasive modality that induces deep neuromuscular activation through rapidly changing magnetic fields, potentially enhancing circulation, muscle recruitment, and neural responsiveness. Although FMS has shown promise in both neurological and musculoskeletal disorders, its combined use with neural mobilization in patients with lumbar radiculopathy has not yet been evaluated in a controlled clinical environment.

Aim: This randomized controlled trial aims to investigate the effectiveness of combining manual therapy with Functional Magnetic Stimulation in adults with chronic lumbar radiculopathy due to lumbar disc herniation. The primary objective is to determine whether the combined intervention provides greater reductions in pain, improved functional capacity, and better neuropathic symptom profiles compared with manual therapy alone.

Method: Forty adults aged 18-64 years with clinically and MRI-confirmed lumbar radiculopathy will be randomly assigned to two groups. The intervention group will participate in a three-week physiotherapy program consisting of manual therapy techniques and Functional Magnetic Stimulation applied 3-4 times per week (10 sessions total). The control group will receive the same manual therapy protocol without FMS. Outcomes will be assessed at baseline and at the end of the three-week intervention period. Primary outcome measures include pain intensity (Numeric Pain Rating Scale, NPRS), functional disability (Roland-Morris Disability Questionnaire, RMDQ), straight leg raise (SLR) angle measured with a goniometer, and neuropathic pain features (S-LANSS, Greek). A mixed-model repeated-measures ANOVA will be used for statistical analysis, with significance set at p < .05.

Expected Results: It is anticipated that individuals receiving the combined manual therapy and FMS intervention will demonstrate greater improvements in pain intensity, functional capacity, and neuropathic symptom characteristics compared with those receiving manual therapy alone.

ELIGIBILITY:
Participants will be eligible for enrollment if they meet all of the following conditions:

* Adults aged 18 to 64 years with a diagnosis of unilateral lumbar disc herniation with radiculopathy (LDHR), established by a spine specialist and confirmed by lumbar MRI demonstrating disc pathology at L4/L5 or L5/S1 impinging on the corresponding nerve root.
* Presence of sciatica-dominant symptoms (radiating pain following the sciatic nerve distribution), accompanied by a positive Straight Leg Raise response consistent with nerve root irritation.
* Symptom duration of at least 12 weeks, indicating a chronic and stable clinical presentation without major fluctuations.
* Referral for physiotherapy management as part of conservative care.
* Ability to comprehend study procedures and provide written informed consent prior to participation.

Exclusion Criteria:

* Candidates will be excluded if any of the following conditions are present:
* Clinical "red flag" indicators such as cauda equina syndrome, suspected spinal infection, or oncologic disease.
* Bilateral radicular involvement or symptoms inconsistent with a single-level LDHR.
* Previous lumbar spine surgery or an upcoming surgical intervention scheduled during the study period.
* Receipt of invasive pain-management procedures (e.g., epidural steroid injections) within the last six weeks.
* Coexisting severe neurologic, metabolic, or inflammatory rheumatologic diseases unrelated to the lumbar radiculopathy.
* Contraindications to magnetic stimulation, including pacemakers, spinal or peripheral neurostimulators, cochlear implants, or clinically significant metallic implants in the stimulation field.
* Pregnancy or breastfeeding.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-11-05 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity with Numeric Rating Scale (NPRS) | pre-treatment, week 3
  Changes in pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), an 11-point scale ranging from 0 to 10. A score of 0 represents "no pain", while 10 represents "the worst possible pain". Two separate pain ratings will be recorded: lumbar pain (NPRS-Lumbar pain) and radicular leg pain (NPRS-Leg pain). Participants will be asked to select the number that best reflects their average pain intensity. The NPRS is a widely accepted tool for evaluating pain in both clinical and research settings, demonstrating excellent test-retest reliability and strong construct validity (Childs et al., 2005).
Straight Leg Raise (SLR) Angle - Goniometry/SROM | pre-treatment, week 3
  Neural mechanosensitivity will be assessed with the passive Straight Leg Raise (SLR) measured using a universal goniometer (SROM). With the participant supine, the hip is passively flexed with the knee extended while the pelvis is stabilized. The assessor records: the Symptom Onset Angle (SOA)-the hip flexion angle (°) at which the participant's typical radicular symptoms first appear. Standardized sensitization maneuvers (e.g., ankle dorsiflexion) may be applied consistently to confirm neural involvement. Higher angles indicate reduced neural mechanosensitivity. The SLR SROM shows good repeatability when the procedure and landmarks are standardized.
Change in Functional Disability | pre-treatment, week 3
  Functional disability will be evaluated using the Roland-Morris Disability Questionnaire (RMDQ), a self-administered instrument specifically designed to measure the impact of low back pain on daily functioning. The questionnaire consists of 24 statements related to physical activities and functional limitations commonly affected by back pain. Participants are asked to mark each statement that applies to them on the day of assessment. The total score ranges from 0 to 24, with higher scores indicating greater disability and reduced functional capacity. The RMDQ is a validated, reliable, and sensitive tool frequently used in both clinical and research contexts to monitor changes in function over time in individuals with low back pain.
Change in Neuropathic Symptom Profile - S-LANSS | pre-treatment, week 3
  Neuropathic pain features will be evaluated with the Self-report Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS), a 7-item questionnaire producing a total score from 0 to 24. Items capture characteristic symptoms (e.g., burning, electric shocks, paresthesias) and symptom behavior. Scores ≥12 suggest pain predominantly of neuropathic origin. The S-LANSS is brief, easy to administer, and has demonstrated acceptable reliability and validity for screening neuropathic pain components and monitoring change over time.

CONTACTS AND LOCATIONS:
Locations (1):
- International Hellenic University, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No